CLINICAL TRIAL: NCT02150018
Title: Effect of Non Invasive Ventilation on Lung Volumes Determined by Electrical Impedance Tomography
Acronym: NIVIT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: University Hospital, Estaing (Other)
Responsible Party: Sponsor
Other Study IDs: CHU-0193
Record Dates: First submitted 2014-05-26; First posted 2014-05-29 (Estimated); Last update posted 2015-07-31 (Estimated); Status verified 2015-07

CONDITIONS: - Critical Care; Non Invasive Ventilation; Electrical Impedance Tomography; End Expiratory Lung Volume; End Expiratory Lung Impedance
Keywords: - Critical Care; Non invasive ventilation; Electrical impedance tomography; End expiratory lung volume; End expiratory lung impedance
MeSH Terms: interventions — Noninvasive Ventilation

STUDY DESIGN:
Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- non invasive ventilation (NIV)
  Interventions: Other: non invasive ventilation

INTERVENTIONS:
Other: non invasive ventilation

SUMMARY:
Effect of Non Invasive Ventilation on end-expiratory lung volumes determined by electrical impedance tomography

DETAILED DESCRIPTION:
Prospective clinical study in ICU with patients requiring non invasive ventilation (NIV) comparing lung volumes determined by electrical impedance tomography before, during and after NIV.

Duration of NIV is 30 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Adult ICU patients requiring non invasive ventilation
* Consent of patients or family
* Arterial line

Exclusion Criteria:

* Tracheotomized patients
* Dressings in the thoracic area

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients requiring non invasive ventilation
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2014-06; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
- End-expiratory lung volume (EELV) determined by electrical impedance tomography before, during and after NIV | at day 1

SECONDARY OUTCOMES:
Anterior, medio-anterior, medio-posterior and posterior EELV | at day 1
Ventilatory frequency | at day 1

CONTACTS AND LOCATIONS:
Overall Officials: Sebastien PERBET, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France